CLINICAL TRIAL: NCT00133055
Title: Parenting Matters: Helping Parents With Young Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Graham J. Reid, Associate Professor, The University of Western Ontario
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67816; 280205-014; ISRCTN81511074
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2011-08

CONDITIONS: Sleep Problems; Behavior Problems; Child Behavior
Keywords: parenting; sleep problems; behavior problems; brief intervention; self-help; preschool-age children; psychosocial
MeSH Terms: conditions — Parasomnias; Mental Disorders; Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Treatment booklet and telephone coaching (Experimental)
  Interventions: Behavioral: Self-help treatment booklet and telephone support
- Usual Care (Other)
  Interventions: Behavioral: Usual care by a family physician

INTERVENTIONS:
Behavioral: Self-help treatment booklet and telephone support — The Parenting Matters treatment program consisted of a self-help treatment booklet and two telephone coaching calls from a paraprofessional telephone coach at Weeks 2 and 5 of the program. Two booklets were used in the three trials; one addressed sleep issues and the second discipline problems.
  Arms: Treatment booklet and telephone coaching
Behavioral: Usual care by a family physician — Parents in the usual care condition were told to continue with care from their family physician and/or any other treatment recommended by the physician.
  Arms: Usual Care

SUMMARY:
Sleep and discipline problems are the most common problems for parents of young children (ages 2 to 5 years old) and are the two concerns with the strongest relations to future child behavior problems. The Parenting Matters program combines treatment booklets and telephone support to help parents deal with sleep or discipline problems. Parents with concerns and who are interested in the study are identified during a visit to their family physician. We, the investigators at the University of Western Ontario, expect that parents receiving treatment booklets, along with usual care by their family physician, will have greater reductions in their child's sleep or discipline problems, improved parenting practices, and greater reductions in child behaviour problems after receiving the Parenting Matters intervention, compared to parents receiving usual medical care.

DETAILED DESCRIPTION:
About 1 in 5 young children (ages 2 to 5 years) has a significant psychosocial problem, but over 80% do not receive treatment. Without treatment, up to half of these children will have problems into childhood and adolescence. New methods of treating and preventing children's psychosocial problems are needed.

Sleep and discipline problems (or child non-compliance) are the most common problems for parents of young children, and are the two concerns with the strongest relations to future child behavior problems. Further, parenting practices have consistently been linked to the development of psychosocial problems. The Parenting Matters program combines treatment booklets and telephone support to help parents with sleep or discipline problems among young children.

Objectives:

* Test the efficacy of the Parenting Matters program interventions for sleeping and bedtime behaviors (Trial 1), and discipline (Trial 2) in reducing problem-specific outcomes.
* Test the effects of the Parenting Matters program interventions for parents who are concerned about both their children's sleep and discipline (Trial 3) in reducing problem-specific outcomes related to sleep (Group 1) and discipline problems (Group 2) will be tested.
* Test the efficacy of the Parenting Matters program in improving parenting practices.
* Test the efficacy of the Parenting Matters program in reducing child behaviour problems in general.
* Examine predictors of treatment success.

Method:

All parents of 2 to 5 year-olds seen in a family practice for a routine appointment are asked to complete a psychosocial concerns checklist. Parents who have concerns regarding their child's sleep (Trial 1), how to discipline their child (Trial 2), or concerns about both their child's sleep and discipline (Trial 3), and meet the other study criteria, are invited to take part in the study. Mailed baseline assessment packages assess children's behavior, parenting practices and potential predictors of treatment success.

Parents are randomized to usual care, or the Parenting Matters program along with usual care. The Parenting Matters program includes treatment booklets addressing either sleep or discipline problems, and telephone coach support (3 calls over 6 weeks).

Primary outcomes are parents' ratings of their children's sleep or discipline problems measured at post-treatment (7 weeks after baseline). Parents repeat assessment packages at 3- and 6-month follow-ups.

Goals & Relevance:

This research addresses the need for new ways of providing early interventions for young children that:

* reach the largest number of individuals in need;
* are cost effective; and
* time efficient.

By addressing the most common issues facing parents of young children, it engages parents in areas of direct relevance to them. The program focuses on parenting practices thereby building family strengths that may have a lasting impact on child development. Collaboration with family physicians builds on the ongoing positive relationships between parents and family physicians and provides a mechanism to reach a significant proportion of young children.

ELIGIBILITY:
Inclusion Criteria:

* Parent (primary caregiver) of a 2-5 year old child
* Attending a medical appointment at a family medical practice
* Phone in home
* Parent concerned about child's sleep and/or discipline
* Parent interested in participating in a treatment study

Exclusion Criteria:

* Parent non-English speaking
* Child with significant physical or developmental disability
* Parent's only sleep concern is in regards to a physiological sleep disorder (e.g. sleep apnea, snoring) or bedwetting
* No phone

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2005-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Sleep and bedtime problems trial (Trial 1): parent report on the Children's Sleep Habits Questionnaire | 7 weeks post randomization
Discipline problems trial (Trial 2): parent rated total problem score on the Eyberg Child Behavior Inventory | 7 weeks post randomization
Sleep and discipline problems trial (Trial 3): parent report on the Children's Sleep Habit Questionnaire (Group 1-sleep treatment) and parent rated total problem score on the Eyberg Child Behavior Inventory (Group 2-discipline treatment) | 7 weeks post randomization

SECONDARY OUTCOMES:
Parenting practices-total score on the Parenting Scale | 7 weeks post randomization; 3- & 6-month follow-up; 12-month follow-up treatment group only
General child behavior problems-total problem score on the Child Behavior Checklist | 7 weeks post randomization; 3- & 6-month follow-up; 12-month follow-up treatment group only
Daily recall ratings of sleep and discipline problems (3 reports in total) | 4 & 6 weeks post randomization; 3- & 6-month follow-up; 12-month follow-up treatment group only
Parent report on the Richman sleep questionnaires (only for Trial 1-sleep and bedtime problems and for Trial 3 participants if in sleep treatment condition) | 7 weeks post randomization; 3- & 6-month follow-up; 12-month follow-up treatment group only

CONTACTS AND LOCATIONS:
Overall Officials: Graham J Reid, PhD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Derived] Reid GJ, Stewart M, Vingilis E, Dozois DJ, Wetmore S, Jordan J, Dickie G, Osmun WE, Wade TJ, Brown JB, Zaric GS. Randomized trial of distance-based treatment for young children with discipline problems seen in primary health care. Fam Pract. 2013 Feb;30(1):14-24. doi: 10.1093/fampra/cms051. Epub 2012 Sep 3. PMID 22948337
- See also: Related Info — http://psychology.uwo.ca/faculty/reid_res.htm